CLINICAL TRIAL: NCT04913311
Title: Predictive Biomarkers for Pneumonitis After Chemoradiotherapy and Immunotherapy
Brief Title: Predictive Biomarkers for Pneumonitis After Chemoradiotherapy and Immunotherapy in Patients With Non-small Cell Lung Cancer
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-0889; NCI-2021-01136 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0889 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-04-20; First posted 2021-06-04 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Lung Non-Small Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Bronchoalveolar Lavage; Bronchoalveolar Lavage Fluid; Chemoradiotherapy; Immune Checkpoint Inhibitors; Nasal Lavage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, stool, saliva, bronchoalveolar lavage and nasal wash sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational (biospecimen collection, standard treatment): Patients undergo collection of blood, stool and saliva samples at baseline. Patients will also have a 6 minute walk and standard of care pulmonary function test at baseline. Patients receive standard of care treatment consisting of concurrent chemoradiation from baseline up to week 10 and immune checkpoint inhibitors from week 10-62. Patients also undergo the collection of blood, stool, saliva and No BAL sample is collected at week 10. During the course of treatment, patients also complete routine tests and procedures to monitor for side effects per standard of care including CT within 4 weeks, lung function tests including home spirometry TIW from week 10-62, bronchoscopy and/or a nasal wash to check for viral infection. Patients also complete questionnaires about symptoms and quality of life QW for weeks 1-10, BIW during weeks 10-62.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bronchoscopy with Bronchoalveolar Lavage; Other: Chemoradiotherapy; Procedure: Computed Tomography; Other: Diagnostic Laboratory Biomarker Analysis; Drug: Immune Checkpoint Inhibitor; Procedure: Nasal Wash and Collection; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Procedure: Spirometry

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood, saliva, stool, and bronchoalveolar lavage samples
Procedure: Bronchoscopy with Bronchoalveolar Lavage — Undergo bronchoscopy with BAL
  Other Names: bronchial washing; Bronchoscopy/Lavage
Other: Chemoradiotherapy — Undergo concurrent chemoradiation per standard of care
  Other Names: Chemoradiation; CRT; CRTx; Radiochemotherapy; RCTx; RT-CT
Procedure: Computed Tomography — Undergo computed tomography scan
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Other: Diagnostic Laboratory Biomarker Analysis — Correlative studies
Drug: Immune Checkpoint Inhibitor — Receive CPI per standard of care
Procedure: Nasal Wash and Collection — Undergo nasal wash
  Other Names: Nasal Lavage; Nasal Wash; Nasopharyngeal Lavage; Nasopharyngeal Wash
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Procedure: Spirometry — Under lung spirometry tests

SUMMARY:
This study looks at the side effects of chemotherapy and radiation (chemoradiation) followed by immunotherapy in patients with non-small cell lung cancer, with a particular focus on lung inflammation (pneumonitis). By collecting blood, stool and saliva samples, and data from lung function tests, researchers may be able to create a database of information about treatment and side effects in patients with non-small cell lung cancer who are receiving chemoradiation followed by immunotherapy. The information gained from this study may also help researchers find signs of problems with lung function earlier rather than later, since lung function is checked more often than routine care. This may improve how quickly these issues can be treated, and future patients may benefit from what is learned.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the association between the incidence of concurrent chemoradiation and subsequent immunotherapy-related adverse events, particularly radiation and immune-related pneumonitis, in patients with non-small cell lung cancer (NSCLC), and various clinicopathologic, radiologic, tumor, and demographic covariates of interest.

SECONDARY OBJECTIVES:

I. To correlate clinicopathologic, radiologic data and tumor characteristics with systemic longitudinal assessments of blood biomarkers for toxicity and response to therapy.

II. To monitor home spirometry and symptoms to identify early pneumonitis. III. To collect blood and microbiome samples from patients on immunotherapy and biopsy samples from toxicity sites at the time of toxicity to evaluate predictive markers for therapy related adverse events.

IV. To determine the effect of concurrent chemotherapy followed by immunotherapy on sleep quality.

V. To determine the impact of sleep disturbance on gut and oral dysbiosis. VI. To characterize longitudinal changes in fatigue and financial toxicity with concurrent chemotherapy followed by immunotherapy.

OUTLINE:

Patients undergo collection of blood, stool and saliva samples at baseline. Patients receive standard of care treatment consisting of concurrent chemoradiation from baseline up to week 62 and immune checkpoint inhibitors from week 10-62. Patients also undergo the collection of blood, stool, saliva and samples at week 10. During the course of treatment, patients also complete routine tests and procedures to monitor for side effects per standard of care including computed tomography (CT) within 4 weeks, lung function tests including home spirometry three times a week (TIW) from week 10-62, bronchoscopy and/or a nasal wash to check for viral infection. Patients also complete questionnaires about symptoms and quality of life once a week (QW) for weeks 1-9, twice a week (BIW) during weeks 5-54, and once a month until week 62.

ELIGIBILITY:
Inclusion Criteria:

* Newly-diagnosed NSCLC patients who will be undergoing concurrent chemotherapy and radiotherapy (XRT) followed by immune checkpoint inhibitors (CPI) therapy with durvalumab, as per the PACIFIC trial
* Willing to undergo all treatment and evaluation at MD Anderson Cancer Center (MDACC)
* Has access to a smartphone with the ability to transmit data via wireless connection or through their personal cellular plan
* Able and willing to perform home spirometry (HS) weekly without absolute contraindications to performing spirometry

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with newly-diagnosed NSCLC (with a particular focus on lung inflammation) scheduled to undergo chemoradiation followed by immunotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-01-21 (Actual); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
Development of pneumonitis during chemoradiotherapy and immunotherapy for locally advanced non-small cell lung cancer (NSCLC) | Up to 12 months
  All possible pneumonitis events will be adjudicated by an expert committee including Dr. Altan, Dr. Sheshadri, an expert infectious disease doctor, and an expert thoracic radiologist. Logistic regression will be used to assess the association between the development of pneumonitis and covariates of interest. Will also use logistic regression to model the association between the development of immune checkpoint inhibitor (CPI)-related pneumonitis and separately the development of radiation related pneumonitis. Secondary analyses of the primary endpoint will include assessing the time to the development of pneumonitis. Cox regression models will be fit in a similar manner to assess the association with the same covariates.

SECONDARY OUTCOMES:
The M.D. Anderson Symptom Index (MDASI) | Up to 12 months
  Monitor home spirometry and symptoms to identify early pneumonitis. The MDASI is a brief (less than 5 minutes), psychometrically validated, multi-symptom assessment tool developed for use with cancer patients who are either undergoing or have completed cancer therapies. MDASI-immunotherapy will be administered weekly for the first 9 weeks of study, every two weeks from week 10 to week 54, and monthly until the end of study (week 62). If MDASI increases by 1, patients will be contacted to be evaluated for the possible development of pneumonitis, infection, or disease progression.
Use of home spirometry | Up to 12 months
  Home spirometry will measured forced lung function values such as vital capacity which will be monitored over time in study participants.
Development of treatment-emergent immune related adverse events (irAE) | Up to 12 months
  The development of treatment-emergent irAE overall and separately by type of AE will be summarized by the method of Kaplan and Meier. For AEs with enough events, may use Cox regression models to model the association with covariates of interest, including blood biomarkers.
Sleep quality | Up to 12 months
  Will assess the association between chemotherapy followed by immunotherapy and sleep quality by using the Pittsburgh Quality Sleep Index (PQSI).
Financial hardship | Up to 12 months
  Will assess the association between financial hardship as measured by changes in the Economic Strain and Resilience in Cancer survey and covariates of interest using linear regression.
Dysbiosis | Up to 12 months
  Will be defined as an abnormal microbiome either measured orally or from the gut bacteria in the stool.

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Sheshadri, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org